CLINICAL TRIAL: NCT04721405
Title: Evaluation of Non-Invasive Assessment for Post RFAL Procedure Monitoring Using the Nanowear Wearable Multiple Sensor Vest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanowear Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NWCT20-SS-003
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Observational Study: No intervention — Observational Study: No intervention

SUMMARY:
The objective of this study is to evaluate an experience of post-operative monitoring using the Nanowear wearable multiple sensor vest in plastic surgery

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* Female and male subjects, at least 18 years of age at the time of enrolment
* The patient is scheduled to undergo BodyTite and/or FaceTite procedures.
* The patients should be willing to comply with the study procedure and schedule.

Exclusion Criteria:

* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* Pregnancy and nursing.
* Subject unwilling or unable to comply with wearing the Nanowear System 12 hours daily for at least 48 hours Up to 7 days
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female over the age of 18 years, healthy adults scheduled to undergo BodyTite and/or FaceTite procedures.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Subject assessment of comfort and compliance | 7 days
  1. Subject assessment of comfort and compliance will be filled out by subjects using a 6-points Usability Survey, as follows:
  * Overall Size of the device - 0 - Being the largest device 5 -Being the smallest.
  * Secrecy - If patient's are uneasy of people knowing they are wearing a medical device. 0 - Not able to hide 5 - Discrete
  * Adaptable to size - Can devices be used on all size patients, extreme scales. 0- Not adjustable 5- Can fit all sizes
  * Device Material - Is the material comfortable to wear. 0 - Uncomfortable 5 - Comfortable
  * Active Wear - Can patient's wear the device while exercising. 0- Not at all 5 - Can exercise without interference.

SECONDARY OUTCOMES:
Investigator assessment of device usability and satisfaction | through study completion, an average of 1 year
  2. Investigator assessment of device usability will be filled out by PI using a 4-points Likert scale, as follows: 3 = Extremely useful in post op care; 2 = Useful in post op care; 1 = Somewhat useful in post op care; 0 = Useless in post op care.
  3. Investigator assessment of satisfaction will be filled out by PI using a 5-points Likert scale, as follows:
  +2 = Very satisfied; +1 = Satisfied; 0 = Indifferent; -1 = Disappointed; -2 = Extremely disappointed.

CONTACTS AND LOCATIONS:
Locations (1):
- Zucker School of Medicine, Hofstra University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No